CLINICAL TRIAL: NCT03213457
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of Elagolix in Combination With Estradiol/Norethindrone Acetate in Subjects With Moderate to Severe Endometriosis-Associated Pain
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Elagolix in Participants With Moderate to Severe Endometriosis-Associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-702
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis
Keywords: Elagolix; Endometriosis associated pain; Dysmenorrhea (DYS); Non-menstrual pelvic pain (NMPP); ORILISSA
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — estradiol, norethindrone drug combination; elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo for elagolix administered twice daily (BID) plus placebo for estradiol/norethindrone acetate (E2/NETA) administered once daily (QD) for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
  Interventions: Drug: Placebo for Elagolix; Drug: Placebo for E2/NETA
- Elagolix / Elagolix + E2/NETA (Experimental): Elagolix 200 mg BID alone for the first 6 months of the 12-month placebo-controlled Treatment Period and elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the second 6 months, followed by elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
  Interventions: Drug: Estradiol/Norethindrone Acetate; Drug: Elagolix
- Elagolix + E2/NETA (Experimental): Elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
  Interventions: Drug: Estradiol/Norethindrone Acetate; Drug: Elagolix

INTERVENTIONS:
Drug: Estradiol/Norethindrone Acetate — Tablets
  Other Names: Activella; E2/NETA
  Arms: Elagolix + E2/NETA; Elagolix / Elagolix + E2/NETA
Drug: Placebo for Elagolix — Tablet
  Arms: Placebo
Drug: Elagolix — Tablet
  Other Names: ABT-620; Elagolix Sodium; ORILISSA
  Arms: Elagolix + E2/NETA; Elagolix / Elagolix + E2/NETA
Drug: Placebo for E2/NETA — Tablets
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate safety and efficacy of elagolix in the management of moderate to severe endometriosis-associated pain in adult premenopausal female participants including the safety and efficacy of elagolix in combination with concomitant hormonal add-back therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a premenopausal female 18 to 49 years of age (inclusive) at the time of Screening.
* Participant has a documented surgical diagnosis (e.g., laparoscopy or laparotomy) of endometriosis established by visualization within 10 years prior to entry into Washout or Screening.
* Participant must agree to use only protocol specified rescue analgesics during the Screening and Treatment Periods for endometriosis-associated pain.
* Participant must have the following documented in the e-Diary during the last 35 days prior to Study Day 1:

  1. At least 2 days of "moderate" or "severe" dysmenorrhea (DYS) AND either
  2. At least 2 days of "moderate" or "severe" non-menstrual pelvic pain (NMPP) and an average NMPP score of at least 1.0, OR
  3. At least 4 days of "moderate" or "severe" NMPP and an average NMPP score of at least 0.5.

Exclusion Criteria:

* Participant has chronic pelvic pain that is not caused by endometriosis, that requires chronic analgesic therapy, which would interfere with the assessment of endometriosis-related pain.
* Participant is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the course of the study. Over-the-counter and prescription topical, inhaled or intranasal corticosteroids are allowed.
* Participant has a history of any major depression or post-traumatic stress disorder (PTSD) within 2 years of the screening visit or other major psychiatric disorder at any time.
* Participant has a history of suicide attempts or answered "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) within the last 1 year at Screening or prior to randomization on Day 1.
* Participant has any history of osteoporosis or other metabolic bone disease or any condition that would interfere with obtaining adequate dual energy x-ray absorptiometry (DXA) measurements
* Screening DXA results of the lumbar spine (L1-L4), femoral neck or total hip bone mineral density (BMD) corresponding to less than 2.0 or more standard deviations below normal.
* Participant has either:

  1. a newly diagnosed, clinically significant medical condition that requires therapeutic intervention (e.g., new onset hypertension), that has not been stabilized 30 days prior to randomization on Day 1 OR
  2. a clinically significant medical condition that is anticipated to require intervention during the course of study participation (e.g., anticipated major elective surgery) OR
  3. an unstable medical condition that makes the subject an unsuitable candidate for the study in the opinion of the Investigator, (including, but not limited to, uncontrolled diabetes mellitus, uncontrolled hypertension, epilepsy requiring anti-epileptic medication, unstable angina, confirmed inflammatory bowel disease, hyperprolactinemia, clinically significant infection or injury).
* Participant has any conditions contraindicated with use of E2/NETA.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 681 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (197):
- United States (188):
  - Central Research Associates /ID# 163087, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC /ID# 145503, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC /ID# 151468, Birmingham, Alabama
  - Southern Women's Specialists PC /ID# 148750, Fairhope, Alabama
  - Women's Health Alliance of Mobile /ID# 150083, Mobile, Alabama
  - University of South Alabama /ID# 148774, Mobile, Alabama
  - Mobile, Ob-Gyn, P.C. /ID# 145364, Mobile, Alabama
  - Mesa Obstetricians and Gynecologists /ID# 147320, Mesa, Arizona
  - Arizona Research Assoc /ID# 161703, Tucson, Arizona
  - Eclipse Clinical Research /ID# 155600, Tucson, Arizona
  - Unity Health- Searcy Medical Center /ID# 203674, Searcy, Arkansas
  - Core Healthcare Group /ID# 149321, Cerritos, California
  - HRC Fertility /ID# 154143, Encino, California
  - Glendale Adventist Medical Ctr /ID# 160530, Glendale, California
  - HCP Clinical Research LLC /ID# 152045, Huntington Beach, California
  - Alliance Research Centers /ID# 151240, Irvine, California
  - Long Beach Clinical Trial Serv /ID# 152428, Long Beach, California
  - Olympia Clinical Trials /ID# 202325, Los Angeles, California
  - California Medical Research As /ID# 154746, Northridge, California
  - Futura Research, Org /ID# 145406, Norwalk, California
  - Huntington Medical Foundation /ID# 154750, Pasadena, California
  - Northern California Research /ID# 159753, Sacramento, California
  - Precision Research Institute - San Diego /ID# 152557, San Diego, California
  - MD Strategies Research Centers /ID# 152429, San Diego, California
  - Alta California Medical Group /ID# 155706, Simi Valley, California
  - Downtown Womens Health Care /ID# 147955, Denver, Colorado
  - Advanced Women's Health Institute /ID# 145396, Greenwood Village, Colorado
  - Red Rocks OB/GYN /ID# 145325, Lakewood, Colorado
  - The Women's Health Group - Thornton /ID# 203707, Thornton, Colorado
  - James A. Simon, MD, PC /ID# 145480, Washington D.C., District of Columbia
  - Helix Biomedics, LLC /ID# 147108, Boynton Beach, Florida
  - Gulf Coast Research Group /ID# 162895, Brandon, Florida
  - Olympian Clinical Research /ID# 148167, Clearwater, Florida
  - Omega Research Maitland, LLC /ID# 145167, DeBary, Florida
  - KO Clinical Research, LLC /ID# 145410, Fort Lauderdale, Florida
  - Clinical Physiology Associates /ID# 145237, Fort Myers, Florida
  - Solutions Through Adv Rch /ID# 148768, Jacksonville, Florida
  - Vida Clinical Research /ID# 150282, Kissimmee, Florida
  - Axcess Medical Center /ID# 148169, Loxahatchee Groves, Florida
  - Genoma Research Group, Inc /ID# 152558, Miami, Florida
  - Vista Health Research LLC - Miami /ID# 151455, Miami, Florida
  - Palmetto Professional Research /ID# 153838, Miami, Florida
  - Precision Research Organization /ID# 145337, Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Inc /ID# 145514, Miami Springs, Florida
  - Salom Tangir, LLC /ID# 148739, Miramar, Florida
  - Suncoast Clinical Research /ID# 145484, New Port Richey, Florida
  - Oncova Clinical Research, Inc. /ID# 148175, Saint Cloud, Florida
  - Physician Care Clin. Res., LLC /ID# 145511, Sarasota, Florida
  - Meridien Research - St Petersburg /ID# 145345, St. Petersburg, Florida
  - Treasure Coast Research /ID# 148174, Stuart, Florida
  - University of South Florida /ID# 145424, Tampa, Florida
  - Stedman Clinical Trials /ID# 152554, Tampa, Florida
  - Virtus Research Consultants, LLC /ID# 147101, Wellington, Florida
  - Comprehensive Clinical Trials /ID# 145148, West Palm Beach, Florida
  - Paramount Research Solutions /ID# 145226, Alpharetta, Georgia
  - Paramount Research Solutions /ID# 149320, Alpharetta, Georgia
  - Agile Clinical Research Trials /ID# 145494, Atlanta, Georgia
  - Atlanta Women's Research Inst /ID# 145543, Atlanta, Georgia
  - Apogee Women's Health Inc. /ID# 145149, College Park, Georgia
  - Columbus Regional Research Ins /ID# 159752, Columbus, Georgia
  - Meridian Clinical Research, LLC /ID# 148176, Savannah, Georgia
  - Atlanta Gynecology Research Institute /ID# 149322, Suwanee, Georgia
  - Clinical Research Prime /ID# 161724, Idaho Falls, Idaho
  - Womens Healthcare Assoc, DBA /ID# 148744, Idaho Falls, Idaho
  - Advanced Clinical Research /ID# 147086, Meridian, Idaho
  - Sonora Clinical Research /ID# 145541, Meridian, Idaho
  - Asr, Llc /Id# 161680, Nampa, Idaho
  - Women's Health Practice, LLC /ID# 145517, Champaign, Illinois
  - Affinity Clinical Research /ID# 151469, Oak Brook, Illinois
  - Center for Women's Research, Inc /ID# 145486, Palos Heights, Illinois
  - The Advanced Gynecologic Surgery Institute - Park Ridge /ID# 151459, Park Ridge, Illinois
  - American Health Network of Ind /ID# 167996, Avon, Indiana
  - Women's Health Advantage /ID# 145495, Fort Wayne, Indiana
  - The Iowa Clinic /ID# 145409, West Des Moines, Iowa
  - Womens & Family Care, LLC dba /ID# 145211, Shawnee Mission, Kansas
  - PRN Professional Research Network of Kansas, LLC /ID# 151463, Wichita, Kansas
  - Cypress Medical Research Ctr /ID# 147159, Wichita, Kansas
  - University of Louisville /ID# 154751, Louisville, Kentucky
  - Bluegrass Clinical Research /ID# 151209, Louisville, Kentucky
  - Clinical Trials Management, LLC - Covington /ID# 145220, Covington, Louisiana
  - Clinical Trials Management, LLC - Covington /ID# 145520, Covington, Louisiana
  - Horizon Research Group /ID# 148171, Eunice, Louisiana
  - Praetorian Pharmaceutical Res /ID# 145405, Marrero, Louisiana
  - Ochsner Baptist OB/GYN Clinic /ID# 147144, New Orleans, Louisiana
  - Women Under Study, LLC /ID# 151216, New Orleans, Louisiana
  - Women's Health Clinic /ID# 155707, Shreveport, Louisiana
  - Omni Fertility and Laser Insti /ID# 145532, Shreveport, Louisiana
  - Eastern Maine Medical Center /ID# 161681, Bangor, Maine
  - Univ Maryland School Medicine /ID# 151739, Baltimore, Maryland
  - Baltimore Suburban Health /ID# 147164, Baltimore, Maryland
  - Continental Clinical Solutions /ID# 152041, Towson, Maryland
  - NECCR Fall River LLC /ID# 145329, Fall River, Massachusetts
  - Genesis Clinical Research - Fall River /ID# 148573, Fall River, Massachusetts
  - ClinSite, LLC /ID# 145314, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc. /ID# 145308, Bay City, Michigan
  - Saginaw Valley Med Res Group /ID# 145527, Saginaw, Michigan
  - Wayne State University Physician Group - Southfield /ID# 145431, Southfield, Michigan
  - Prism Research /ID# 159751, Saint Paul, Minnesota
  - Womens Clinic of Lincoln, P.C. /ID# 145366, Lincoln, Nebraska
  - Accent Clinical Trials /ID# 147109, Las Vegas, Nevada
  - Office of Edmond E. Pack, MD /ID# 148747, Las Vegas, Nevada
  - R. Garn Mabey Jr, MD Chartered /ID# 145361, Las Vegas, Nevada
  - Jersey Shore University Medical Center /ID# 148756, Neptune City, New Jersey
  - Rutgers Robert Wood Johnson /ID# 152858, New Brunswick, New Jersey
  - St. Joseph's Regional Medical /ID# 157759, Totowa, New Jersey
  - Albuquerque Clinical Trials, Inc /ID# 154747, Albuquerque, New Mexico
  - Bosque Women's Care /ID# 147084, Albuquerque, New Mexico
  - SUNY Downstate Medical Center /ID# 148749, Brooklyn, New York
  - Scott Research Inc. /ID# 161704, Laurelton, New York
  - Manhattan Medical Research /ID# 145175, New York, New York
  - Columbia Univ Medical Center /ID# 145334, New York, New York
  - Hamburg Regional Gynecology Gr /ID# 161705, Orchard Park, New York
  - OB.GYN Associates of WNY /ID# 161665, West Seneca, New York
  - PMG Research of Charlotte /ID# 145432, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 154679, Charlotte, North Carolina
  - Carolina Women's Research and Wellness Center /ID# 145356, Durham, North Carolina
  - Unified Women's Clinical Research-Greensboro /ID# 155543, Greensboro, North Carolina
  - Pinewest Ob-Gyn, Inc. /ID# 151743, High Point, North Carolina
  - Eastern Carolina Women's Centr /ID# 145386, New Bern, North Carolina
  - Unified Women's Clinical Resea /ID# 145353, Raleigh, North Carolina
  - PMG Research of Wilmington /ID# 152555, Wilmington, North Carolina
  - Trinity Health Center Town /ID# 147102, Minot, North Dakota
  - Clinical Inquest Center Ltd /ID# 147107, Beavercreek, Ohio
  - CTI Clinical Research Center /ID# 145428, Cincinnati, Ohio
  - The Christ Hospital /ID# 149244, Cincinnati, Ohio
  - University of Cincinnati /ID# 145496, Cincinnati, Ohio
  - Univ Hosp Cleveland /ID# 148741, Cleveland, Ohio
  - The Ohio State University /ID# 145444, Columbus, Ohio
  - Aventiv Research, Inc. /ID# 145492, Columbus, Ohio
  - Aventiv Research, Inc. /ID# 162896, Columbus, Ohio
  - Wright State University & CTRA /ID# 145512, Fairborn, Ohio
  - University of Toledo /ID# 145403, Toledo, Ohio
  - Oregon Health and Science University /ID# 155705, Portland, Oregon
  - Main Line Fertility Center /ID# 150099, Bryn Mawr, Pennsylvania
  - OB/GYN Associates of Erie /ID# 157935, Erie, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 145231, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 145470, Philadelphia, Pennsylvania
  - Drexel Univ College of Med /ID# 149789, Philadelphia, Pennsylvania
  - Frontier Clinical Research /ID# 162091, Smithfield, Pennsylvania
  - Vista Clinical Research /ID# 148767, Columbia, South Carolina
  - University Medical Group /ID# 148777, Greenville, South Carolina
  - Venus Gynecology, LLC /ID# 145336, Myrtle Beach, South Carolina
  - James T. Martin, Jr., MD., Obs /ID# 148755, North Charleston, South Carolina
  - Palmetto Clinical Research /ID# 150992, Summerville, South Carolina
  - Brown Clinic, PLLP /ID# 154372, Watertown, South Dakota
  - Holston Medical Group /ID# 145449, Bristol, Tennessee
  - Chattanooga Medical Research /ID# 145184, Chattanooga, Tennessee
  - WR-ClinSearch /ID# 145205, Chattanooga, Tennessee
  - The Jackson Clinic, PA /ID# 145303, Jackson, Tennessee
  - Research Memphis Associates, LLC /ID# 150100, Memphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 145224, Nashville, Tennessee
  - Lotus Gynecology /ID# 148479, Austin, Texas
  - AA (Austin Area) ObGyn PLLC /ID# 205696, Austin, Texas
  - Sirius Clinical Research, LLC /ID# 154749, Austin, Texas
  - Gadolin Research, LLC /ID# 201383, Beaumont, Texas
  - Center for Assisted Reprod. /ID# 154748, Bedford, Texas
  - Texas Health Presbyterian Hosp /ID# 150098, Dallas, Texas
  - UT Southwestern Medical Center /ID# 145201, Dallas, Texas
  - Baylor Scott & White /ID# 170430, Fort Worth, Texas
  - Signature Gyn Services /ID# 145534, Fort Worth, Texas
  - Willowbend Health and Wellness - Frisco /ID# 145245, Frisco, Texas
  - Next Innovative Clinical Research /ID# 203863, Houston, Texas
  - Advances in Health, Inc. /ID# 145425, Houston, Texas
  - Houston Methodist Hospital /ID# 170586, Houston, Texas
  - Precision Research Institute - Houston /ID# 154370, Houston, Texas
  - The Woman's Hospital of Texas /ID# 145316, Houston, Texas
  - Centex Studies, Inc /ID# 148776, Houston, Texas
  - FMC Science /ID# 150981, Lampasas, Texas
  - Clinical Trials of Texas, Inc /ID# 147100, San Antonio, Texas
  - VIP Trials /ID# 151745, San Antonio, Texas
  - Discovery Clinical Trials-San Antonio /ID# 145363, San Antonio, Texas
  - Houston Ctr for Clin Research /ID# 148799, Sugar Land, Texas
  - Center of Reproductive Medicin /ID# 145467, Webster, Texas
  - Corner Canyon Obstetrics and G /ID# 145519, Draper, Utah
  - Tanner Clinic /ID# 148786, Layton, Utah
  - Revere Health /ID# 145540, Pleasant Grove, Utah
  - Southampton Women's Health /ID# 151691, Franklin, Virginia
  - Health Research of Hampton Roads, Inc. (HRHR) /ID# 156477, Newport News, Virginia
  - Clinical Research Partners, LL /ID# 145392, North Chesterfield, Virginia
  - Clinical Research Partners, LL /ID# 145416, North Chesterfield, Virginia
  - Clinical Trials Virginia, Inc. /ID# 145430, Richmond, Virginia
  - Alliance Womens Health /ID# 148770, Richmond, Virginia
  - Tidewater Clinical Research /ID# 145397, Virginia Beach, Virginia
  - Clinical Research Adv, Inc. /ID# 149257, Puyallup, Washington
  - Virginia Mason Medical Center /ID# 145387, Seattle, Washington
  - Seattle Women's Health, Research, Gynecology /ID# 145341, Seattle, Washington
  - North Spokane Women's Health /ID# 145382, Spokane, Washington
  - Madigan Army Medical Center /ID# 145186, Tacoma, Washington
- Canada (5):
  - Strand Clinic /ID# 152582, St. John's, Newfoundland and Labrador
  - Medicor Research Inc /ID# 151453, Greater Sudbury, Ontario
  - The Ottawa Hospital /ID# 148927, Ottawa, Ontario
  - Mount Sinai Hosp.-Toronto /ID# 148972, Toronto, Ontario
  - Victory Reproductive Care /ID# 149016, Windsor, Ontario
- Puerto Rico (4):
  - Puerto Rico Medical Research /ID# 152040, Ponce
  - Clinical Research Puerto Rico /ID# 149018, San Juan
  - Rodriguez-Ginorio, San Juan /ID# 145545, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 145546, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Watts NB, Binkley N, Owens CD, Al-Hendy A, Puscheck EE, Shebley M, Schlaff WD, Simon JA. Bone Mineral Density Changes Associated With Pregnancy, Lactation, and Medical Treatments in Premenopausal Women and Effects Later in Life. J Womens Health (Larchmt). 2021 Oct;30(10):1416-1430. doi: 10.1089/jwh.2020.8989. Epub 2021 Aug 25. PMID 34435897
- See also: Related info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 679 subjects were treated at 137 sites in 2 countries (US [including Puerto Rico] and Canada). Of the 679 subjects who were treated on study, 299 subjects discontinued study drug prematurely during the Placebo-Controlled Treatment Period and 240 discontinued study drug prematurely during the Open-Label Treatment Period.
Pre-assignment Details: Participants were randomly assigned on Study Day 1 in a 4:1:2 ratio as follows:
  * elagolix 200 mg twice daily (BID) plus estradiol/norethindrone acetate (E2/NETA) 1 mg/0.5 mg once daily (QD)
  * elagolix 200 mg BID
  * placebo
  Data are presented for the 12-month Placebo-Controlled Treatment Period.
Groups:
- Placebo: Placebo for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- Elagolix / Elagolix + E2/NETA: Elagolix 200 mg BID alone for the first 6 months of the 12-month placebo-controlled Treatment Period and elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the second 6 months, followed by elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
Period: Screening Period
Arm/Group | Placebo | Elagolix / Elagolix + E2/NETA | Elagolix + E2/NETA
Started (Includes all randomized participants.) | 194 | 98 | 389
Completed | 193 | 97 | 389
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0
Period: Double-Blind Period
Arm/Group | Placebo | Elagolix / Elagolix + E2/NETA | Elagolix + E2/NETA
Started (Includes all treated participants who received at least one dose of study drug.) | 193 | 97 | 389
Completed | 157 | 85 | 337
Not Completed | 36 | 12 | 52
Not completed — Adverse Event | 3 | 2 | 7
Not completed — Withdrawal by Subject | 14 | 2 | 14
Not completed — Lost to Follow-up | 2 | 3 | 9
Not completed — Requires surgery or invasive intervention for treatment of endometriosis | 2 | 0 | 1
Not completed — Non-compliance with study procedures | 0 | 2 | 4
Not completed — Pregnancy | 5 | 0 | 0
Not completed — Other | 10 | 3 | 17
Period: Open-Label Period
Arm/Group | Placebo | Elagolix / Elagolix + E2/NETA | Elagolix + E2/NETA
Started (Includes participants who completed the Placebo-Controlled Treatment Period and entered the Open-Label Treatment Period.) | 106 | 59 | 215
Completed | 90 | 48 | 170
Not Completed | 16 | 11 | 45
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Withdrawal by Subject | 12 | 5 | 24
Not completed — Lost to Follow-up | 1 | 2 | 8
Not completed — Requires surgery or invasive intervention for treatment of endometriosis | 0 | 0 | 2
Not completed — Non-compliance with study procedures | 1 | 1 | 2
Not completed — Exclusionary medications | 0 | 0 | 1
Not completed — Other | 1 | 1 | 6
Period: Follow-Up Period
Arm/Group | Placebo | Elagolix / Elagolix + E2/NETA | Elagolix + E2/NETA
Started (Includes all randomized participants. Participants were expected to enter the Follow-Up Period after Treatment Month 48, or if a participant prematurely discontinued from the Treatment Period at the time of or after Treatment Month 6.) | 194 | 98 | 389
Completed | 102 | 51 | 185
Not Completed | 92 | 47 | 204
Not completed — Adverse Event | 16 | 8 | 37
Not completed — Withdrawal by Subject | 18 | 11 | 55
Not completed — Lost to Follow-up | 28 | 15 | 50
Not completed — Requires surgery or invasive intervention for treatment of endometriosis | 3 | 1 | 2
Not completed — Non-compliance with study procedures | 4 | 1 | 6
Not completed — Pregnancy | 7 | 0 | 18
Not completed — Exclusionary medications | 1 | 1 | 5
Not completed — COVID-19 logistical restrictions | 1 | 0 | 0
Not completed — Other | 14 | 10 | 31

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix / Elagolix + E2/NETA | Elagolix + E2/NETA | Total
Number analyzed (Participants) | 193 | 97 | 389 | 679
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (6.72) | 32.5 (6.44) | 32.3 (6.74) | 32.5 (6.69)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 193 | 97 | 389 | 679
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 11 | 58 | 106
  Not Hispanic or Latino | 156 | 86 | 331 | 573
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 31 | 19 | 49 | 99
  White | 159 | 74 | 328 | 561
  More than one race | 2 | 4 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Endpoint: Percentage of Participants With a Response for Dysmenorrhea (DYS) at Months 6 and 12 Based on Daily Assessment
Description: Participants recorded rescue analgesic use for endometriosis-associated pain daily and DYS (pain during menstruation ) and its impact on daily activities each day of their period in an electronic diary (e-Diary). DYS was measured by the 4-point Endometriosis Daily Pain Impact Diary according to the following:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores and analgesic use were averaged over 35 days prior to each visit.
  Response was defined as a reduction of -0.92 or more from baseline in DYS as well as no increase in rescue analgesic use for endometriosis-associated pain (defined as a < 15% increase in average rescue analgesic pill count and no additional analgesic).
Time Frame: Month 6, Month 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants with an assessment at given time point. Last observation carried forward. Per protocol, the primary comparison for the co-primary endpoints was between the elagolix plus E2/NETA and placebo arms only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 190 | 384
percentage of participants
  Month 6 | 23.7 [17.64 to 29.73] | 62.8 [57.93 to 67.60]
  Month 12: number analyzed (Participants) | 189 | 376
  Month 12 | 29.1 [22.62 to 35.58] | 63.8 [58.97 to 68.69]
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — P-value for test of difference is from a logistic regression model including treatment as the main effect and baseline value as a covariate; Odds Ratio (OR) = 5.51, 95% CI 2-sided [3.711 to 8.176]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Month 12; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.33, 95% CI 2-sided [2.968 to 6.331]

2. Primary Outcome: Co-Primary Endpoint: Percentage of Participants With a Response for Non-menstrual Pelvic Pain (NMPP) at Months 6 and 12 Based on Daily Assessment
Description: Participants recorded rescue analgesic medication for endometriosis-associated pain and assessed NMPP and its impact on their daily activities each day in an e-Diary was measured by the 4-point Endometriosis Daily Pain Impact Diary according to the following:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores and analgesic use were averaged over the 35 days prior to each visit.
  Response was defined as a reduction of -0.55 or greater from baseline for NMPP as well as no increase in rescue analgesic use for endometriosis-associated pain (defined as a < 15% increase in average pill count of rescue analgesics and no additional analgesics).
Time Frame: Month 6, Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 190 | 384
percentage of participants
  Month 6 | 36.8 [29.98 to 43.70] | 51.3 [46.30 to 56.30]
  Month 12: number analyzed (Participants) | 189 | 376
  Month 12 | 42.3 [35.28 to 49.37] | 54.3 [49.22 to 59.29]
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.275 to 2.605]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Month 12; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.146 to 2.326]

3. Secondary Outcome: Change From Baseline in DYS at Month 12 Based on Daily Assessment
Description: Participants assessed DYS (pain during menstruation) and its impact on their daily activities each day of their period in an e-Diary. DYS was measured by the 4-point Endometriosis Daily Pain Impact Diary according to the following:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores were averaged over the 35 days prior to each visit.
Time Frame: Baseline, Month 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants with an assessment. Mixed-effects model repeated measures (MMRM) analysis. Per protocol, the primary comparison for the secondary endpoints was between the elagolix plus E2/NETA and placebo arms only.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 111 | 216
score on a scale | -0.73 (0.077) | -1.73 (0.055)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; Ranked secondary endpoints were tested following a fixed-sequence testing procedure. Testing began with testing each of the co-primary endpoints using alpha of 0.05 (2-sided) for elagolix plus E2/NETA compared to placebo. If both co-primary endpoints achieved statistical significance with elagolix plus E2/NETA as compared to placebo, continued testing was performed for the ranked secondary endpoints following a fixed-sequence testing procedure in the order of endpoints presented; Test type: Superiority; p < 0.001, mixed model repeated measures (MMRM) — P value for the test of the difference is from an MMRM with the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, and the continuous fixed covariate of baseline pain score, and random effect for participant; Least Squares (LS) Mean of Difference = -0.99, 95% CI 2-sided [-1.180 to -0.809], Standard Error of Mean 0.094

4. Secondary Outcome: Change From Baseline in DYS at Month 6 Based on Daily Assessment
Description: Participants assessed DYS (pain during menstruation) and its impact on their daily activities each day of their period in an e-Diary. DYS was measured by the 4-point Endometriosis Daily Pain Impact Diary according to the following:
  0: No discomfort
  1. Mild discomfort but I was easily able to do the things I usually do
  2. Moderate discomfort or pain that made it difficult to do some of the things I usually do
  3. Severe pain that made it difficult to do the things I usually do.
  Pain scores were averaged over the 35 days prior to each visit.
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 138 | 286
score on a scale | -0.62 (0.072) | -1.64 (0.050)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.02, 95% CI 2-sided [-1.190 to -0.845], Standard Error of Mean 0.088

5. Secondary Outcome: Change From Baseline in DYS at Month 3 Based on Daily Assessment
Description: as for outcome 4
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 170 | 335
score on a scale | -0.56 (0.069) | -1.54 (0.049)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.99, 95% CI 2-sided [-1.156 to -0.823], Standard Error of Mean 0.085

6. Secondary Outcome: Change From Baseline in Non-menstrual Pelvic Pain (NMPP) at Month 12 Based on Daily Assessment
Description: Participants recorded rescue analgesic medication for endometriosis-associated pain and assessed NMPP and its impact on their daily activities each day in an e-Diary was measured by the 4-point Endometriosis Daily Pain Impact Diary according to the following:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores and analgesic use were averaged over the 35 days prior to each visit.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 111 | 216
score on a scale | -0.64 (0.060) | -0.86 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.22, 95% CI 2-sided [-0.367 to -0.080], Standard Error of Mean 0.073

7. Secondary Outcome: Change From Baseline in NMPP at Month 6 Based on Daily Assessment
Description: as for outcome 6
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 138 | 286
score on a scale | -0.57 (0.051) | -0.78 (0.036)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.21, 95% CI 2-sided [-0.329 to -0.085], Standard Error of Mean 0.062

8. Secondary Outcome: Change From Baseline in NMPP at Month 3 Based on Daily Assessment
Description: as for outcome 6
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 170 | 335
score on a scale | -0.49 (0.046) | -0.65 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.16, 95% CI 2-sided [-0.270 to -0.050], Standard Error of Mean 0.056

9. Secondary Outcome: Change From Baseline to Month 6 in Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Short Form 6a T-Score
Description: The PROMIS Fatigue Short Form 6a is self-administered and composed of 6 questions to evaluate fatigue over the past 7 days. All questions employ the following five response options: 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, and 5 = Always. The PROMIS Fatigue 6a score is calculated as a T-score, which is a standardized score with a mean of 50 (based on the average for the United States general population) and a standard deviation (SD) of 10. Higher scores indicate higher levels of fatigue. A decrease in score (negative change from baseline) indicates improvement in fatigue.
Time Frame: Baseline, Month 6
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants with an assessment. Observed cases. Per protocol, the primary comparison for the secondary endpoints was between the elagolix plus E2/NETA and placebo arms only.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 146 | 302
T-score | -4.71 (0.739) | -7.22 (0.514)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.005, ANCOVA — P-value for test of difference at each post-baseline time point is from an ANCOVA model with treatment as the main effect and baseline as a covariate; LS Mean of Difference = -2.51, 95% CI 2-sided [-4.283 to -0.746], Standard Error of Mean 0.900

10. Secondary Outcome: Change From Baseline in Dyspareunia (DYSP) at Month 12 Based on Daily Assessment
Description: Participants assessed DYSP each day in an e-Diary according to the following response options:
  * 0: None; No discomfort during sexual intercourse
  * 1: Mild; Able to tolerate the discomfort during sexual intercourse
  * 2: Moderate; Intercourse was interrupted due to pain
  * 3: Severe; Avoided intercourse because of pain
  * Not applicable; I was not sexually active for reasons other than endometriosis or did not have sexual intercourse.
  Pain scores were averaged over the 35 days prior to each visit. Responses of "Not Applicable" were excluded.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 84 | 147
score on a scale | -0.60 (0.079) | -0.70 (0.058)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.284, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.298 to 0.088], Standard Error of Mean 0.098

11. Secondary Outcome: Change From Baseline in DYSP at Month 6 Based on Daily Assessment
Description: as for outcome 10
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 96 | 209
score on a scale | -0.54 (0.076) | -0.63 (0.053)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.286, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.10, 95% CI 2-sided [-0.279 to 0.083], Standard Error of Mean 0.092

12. Secondary Outcome: Change From Baseline in DYSP at Month 3 Based on Daily Assessment
Description: as for outcome 10
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 119 | 257
score on a scale | -0.40 (0.064) | -0.62 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; Ranked secondary endpoints were tested following a fixed-sequence testing procedure. Testing began with testing each of the co-primary endpoints using alpha of 0.05 (2-sided) for elagolix plus E2/NETA compared to placebo. If both co-primary endpoints achieved statistical significance with elagolix E2/NETA as compared to placebo, continued testing was performed for the ranked secondary endpoints following a fixed-sequence testing procedure in the order of endpoints presented; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.22, 95% CI 2-sided [-0.375 to -0.066], Standard Error of Mean 0.079

13. Secondary Outcome: Change From Baseline to Month 12 in Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Short Form 6a T-Score
Description: as for outcome 9
Time Frame: Baseline, Month 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 108 | 220
T-score | -6.43 (0.949) | -8.92 (0.665)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.032, ANCOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean of Difference = -2.49, 95% CI 2-sided [-4.773 to -0.216], Standard Error of Mean 1.158

14. Secondary Outcome: Change From Baseline in Endometriosis-Associated Pain Score at Month 12 Assessed With Numeric Rating Scale (NRS)
Description: The NRS measured endometriosis-associated pain with and without menstruation on an 11-point scale from 0 = no pain to 10 = worst pain ever. Site staff administered the Overall Endometriosis-Associated Pain questionnaire assessing pain over a 7-day recall period, and recorded the participant's response electronically via a tablet at the time of visit. Pain scores were averaged over the 35 days prior to each visit.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 102 | 202
score on a scale | -3.25 (0.263) | -4.39 (0.186)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.14, 95% CI 2-sided [-1.774 to -0.508], Standard Error of Mean 0.322

15. Secondary Outcome: Change From Baseline in Endometriosis-Associated Pain Score at Month 6 Assessed With NRS
Description: as for outcome 14
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 130 | 269
score on a scale | -2.74 (0.248) | -4.12 (0.174)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.38, 95% CI 2-sided [-1.978 to -0.788], Standard Error of Mean 0.303

16. Secondary Outcome: Change From Baseline in Endometriosis-Associated Pain Score at Month 3 Assessed With NRS
Description: as for outcome 14
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Elagolix + E2/NETA: Elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA [1 mg/0.5 mg] QD for the remaining 36 months of the Treatment Period.
Arm/Group | Placebo | Elagolix + E2/NETA
Number analyzed (Participants) | 156 | 304
score on a scale | -2.33 (0.225) | -3.79 (0.161)
Statistical Analysis 1: Comparison: Placebo vs Elagolix + E2/NETA; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.46, 95% CI 2-sided [-2.002 to -0.915], Standard Error of Mean 0.276

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization through the end of the Treatment Period (Month 12). Adverse Events(AEs): From first dose of study drug through the end of the Treatment Period (Month 12).
Description: Treatment emergent AEs (TEAEs) during the 12-Month Placebo-Controlled Treatment Period are presented, and are defined as those that occurred no more than 30 days after the last dose of study drug for participants who discontinued prematurely or until the first dose of the study drug in the Open-Label Treatment.
  Arm counts include all randomized participants.
Groups:
- SCR_Placebo: Screening (SCR) Period: Placebo for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- SCR_Elagolix: Screening (SCR) Period: Elagolix 200 mg BID alone for the first 6 months of the 12-month placebo-controlled Treatment Period and elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the second 6 months, followed by elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- SCR_Elagolix_and_E2-NETA: Screening (SCR) Period: Elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- DB_Placebo: Double-blinded (DB) Period: Placebo for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- DB_Elagolix: Double-blinded (DB) Period: Elagolix 200 mg BID alone for the first 6 months of the 12-month placebo-controlled Treatment Period and elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the second 6 months, followed by elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- DB_Elagolix_and_E2-NETA: Double-blinded (DB) Period: Elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- OL_Placebo_to_ELA_and_E2-NETA: Open-Label (OL) Period: Placebo for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- OL_ELA_to_ELA_and_E2-NETA: Open-Label (OL) Period: Elagolix 200 mg BID alone for the first 6 months of the 12-month placebo-controlled Treatment Period and elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the second 6 months, followed by elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- OL_ELA_and_E2-NETA_to_ELA_and_E2-NETA: Open-Label (OL) Period: Elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- FU_Placebo_to_ELA_and_E2-NETA: Follow-Up (FU) Period: Placebo for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- FU_ELA_to_ELA_and_E2-NETA: Follow-Up (FU) Period: Elagolix 200 mg BID alone for the first 6 months of the 12-month placebo-controlled Treatment Period and elagolix 200 mg BID+E2/NETA 1 mg/0.5 mg QD for the second 6 months, followed by elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
- FU_ELA_and_E2-NETA_to_ELA_and_E2-NETA: Follow-Up (FU) Period: Elagolix 200 mg BID + E2/NETA 1 mg/0.5 mg QD for the 12-month placebo-controlled Treatment Period, followed by elagolix 200 mg BID plus E2/NETA 1 mg/0.5 mg QD for the remaining 36 months of the Treatment Period.
Arm/Group | SCR_Placebo | SCR_Elagolix | SCR_Elagolix_and_E2-NETA | DB_Placebo | DB_Elagolix | DB_Elagolix_and_E2-NETA | OL_Placebo_to_ELA_and_E2-NETA | OL_ELA_to_ELA_and_E2-NETA | OL_ELA_and_E2-NETA_to_ELA_and_E2-NETA | FU_Placebo_to_ELA_and_E2-NETA | FU_ELA_to_ELA_and_E2-NETA | FU_ELA_and_E2-NETA_to_ELA_and_E2-NETA
All-Cause Mortality (participants affected / at risk) | 0/194 | 0/98 | 0/389 | 0/194 | 0/98 | 0/389 | 0/106 | 0/59 | 0/215 | 0/194 | 0/98 | 0/389
Serious Adverse Events (participants affected / at risk) | 0/194 | 0/98 | 1/389 | 8/194 | 2/98 | 14/389 | 7/106 | 2/59 | 10/215 | 2/194 | 0/98 | 1/389
Other Adverse Events (participants affected / at risk) | 1/194 | 0/98 | 1/389 | 89/194 | 74/98 | 236/389 | 60/106 | 32/59 | 125/215 | 2/194 | 3/98 | 6/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCR_Placebo (N=194) | SCR_Elagolix (N=98) | SCR_Elagolix_and_E2-NETA (N=389) | DB_Placebo (N=194) | DB_Elagolix (N=98) | DB_Elagolix_and_E2-NETA (N=389) | OL_Placebo_to_ELA_and_E2-NETA (N=106) | OL_ELA_to_ELA_and_E2-NETA (N=59) | OL_ELA_and_E2-NETA_to_ELA_and_E2-NETA (N=215) | FU_Placebo_to_ELA_and_E2-NETA (N=194) | FU_ELA_to_ELA_and_E2-NETA (N=98) | FU_ELA_and_E2-NETA_to_ELA_and_E2-NETA (N=389)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PITUITARY APOPLEXY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PITUITARY TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VESTIBULAR MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVICAL INCOMPETENCE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCR_Placebo (N=194) | SCR_Elagolix (N=98) | SCR_Elagolix_and_E2-NETA (N=389) | DB_Placebo (N=194) | DB_Elagolix (N=98) | DB_Elagolix_and_E2-NETA (N=389) | OL_Placebo_to_ELA_and_E2-NETA (N=106) | OL_ELA_to_ELA_and_E2-NETA (N=59) | OL_ELA_and_E2-NETA_to_ELA_and_E2-NETA (N=215) | FU_Placebo_to_ELA_and_E2-NETA (N=194) | FU_ELA_to_ELA_and_E2-NETA (N=98) | FU_ELA_and_E2-NETA_to_ELA_and_E2-NETA (N=389)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 12 (12) | 16 (19) | 51 (55) | 9 (11) | 2 (3) | 12 (13) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 17 (17) | 1 (1) | 4 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 11 (11) | 5 (5) | 6 (7) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 7 (8) | 29 (32) | 1 (1) | 0 (0) | 2 (2)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 9 (9) | 2 (2) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 9 (9) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 4 (4) | 16 (16) | 3 (3) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 5 (5) | 21 (24) | 2 (3) | 3 (3) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 10 (10) | 32 (34) | 9 (13) | 5 (5) | 18 (28) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 7 (8) | 17 (18) | 6 (6) | 1 (2) | 13 (15) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 9 (10) | 15 (15) | 6 (7) | 5 (7) | 16 (19) | 1 (1) | 1 (1) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 16 (21) | 3 (4) | 4 (5) | 14 (18) | 0 (0) | 0 (0) | 0 (0)
BONE DENSITY DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 7 (7) | 6 (6) | 21 (21) | 0 (0) | 1 (1) | 1 (1)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 2 (2) | 7 (7) | 4 (5) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (6) | 15 (17) | 6 (6) | 3 (7) | 8 (8) | 0 (0) | 1 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 22 (22) | 2 (2) | 2 (3) | 15 (17) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 10 (10) | 13 (13) | 46 (47) | 8 (9) | 4 (5) | 7 (8) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 19 (24) | 6 (6) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 18 (18) | 7 (7) | 3 (3) | 17 (20) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 12 (13) | 2 (3) | 2 (2) | 15 (18) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 13 (15) | 5 (5) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
MOOD SWINGS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 21 (21) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (8) | 18 (20) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 17 (17) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 13 (14) | 24 (25) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 14 (15) | 43 (44) | 69 (74) | 8 (9) | 2 (2) | 10 (11) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03213457/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03213457/SAP_001.pdf